CLINICAL TRIAL: NCT04324177
Title: Profile and Clinical Outcome of Pediatric Patients Admitted to Intensive Care Unit of Assiut University Children Hospital
Brief Title: Profile of Pediatric Patients Admitted to AU ICU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, GM Abdelsalam, Principal investigator, Assiut University
Other Study IDs: gehad011157
Record Dates: First submitted 2020-03-19; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Demography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Demographic data, morbidity data — To detect association between the demographic data of pediatric patients including age ,sex,hospital stay and clinical data including the diagnosis and co morbidity with the outcome of pediatric patients admitted to ICU of Assiut University children hospital

SUMMARY:
This study aims to determine the profile and outcome of children admitted to ICU at Assiut University children hospital in order to detect association between risk factors and outcome, to asses the efficacy of treatment making it possible to take better decisions , to improve the quality of care.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to intensive care unit of Assiut University children hospital over one year aged from 1month to 18 years

Exclusion Criteria:

* pediatric patients less than one month old Pediatric patients will die on arrival

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All patients admitted to the PICU whichever is the diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients according to age groups and gender | 1 year
  The demographic data (including age groups and gender).
  Regarding age groups, the number of patients in each of three groups will be addressed:
  1. 1 month to 2 years of age
  2. 2 years to 12 years of age
  3. 12 to 18 years of age"
  Regarding gender, the number of patients will be allocated in 2 groups:
  1. male
  2. female
Number of patients according to diagnosis on admission | 1 year
  Provisional diagnosis on admission categorised by the system affected (respiratory, cardiovascular, neurological, hematological, renal, endocrinal and metabolic gastrointestinal and hepatobiliary, multi system affection, others (post operative, post arrest, sepsis syndrome, malignancies, poisoning, coma of unknownorigin)). The data will be presented as number of patients in each group of system affected.
Number of patients according to referral site | 1 year
  The patients will be allocated in 2 groups of referral sites of patients admitted to the PICU:
  1. the ward
  2. the emergency department. Data will be presented as number of patients in each group.
Number of patients according to the need for mechanical ventilation and its duration | 1 year
  The patients will be allocated in 2 groups based on the need for mechanical ventilation duringthe PICU stay. In case of need for mechanical ventilation, the duration will be recorded in days.
Length of stay in days | 1 year
  Length of stay in the pediatric intensive care unit (PICU) will be presented as number of days spent by the patient from admission to discharge or death.
Pediatric Risk of Mortality score on admission | 1 year
  Pediatric Risk of Mortlaity (PRISM) III score will be obtained from all patients within the first 24 hours of admission to the PICU. The maximum total PRISM III score is 74. The higher the score, the worse the prognosis. For the analysis of mortality risk factors, patients will be allocated into two groups according to PRISM III 24 score values >8 and ≤ 8, based on previously published data showing increased mortality risk in patients with PRISM III 24 score >8.
Number of patients according to the condition of discharge from the pediatric intensive care unit | 1 year
  Number of patients discharged from the PICU allocated in 2 groups:
  1. improvent and transfer to the corresponding medical ward. (Survivors)
  2. death. N.B. patients who will be discharged against medical advice (DAMA) will be excluded from the proposed data analysis, but will be pointed at.

SECONDARY OUTCOMES:
Correlation 1 | 1 year
  Correlation between number of patients in discharge groups (survivors / dead) and age group.
Correlation 2 | 1 year
  Correlation between number of patients in discharge groups (survivors / dead) and diagnosis on admission.
Correlation 3 | 1 year
  Correlation between number of patients in discharge groups (survivors / dead) and length of stay.
Correlation 4 | 1 year
  Correlation between number of patients in discharge groups (survivors / dead) and PRISM III score.
Correlation 5 | 1 year
  Correlation between number of patients in discharge groups (survivors / dead) and duration of mechanical ventilation.

REFERENCES:
- [Background] Haftu H, Hailu T, Medhaniye A, G/Tsadik T. Assessment of pattern and treatment outcome of patients admitted to pediatric intensive care unit, Ayder Referral Hospital, Tigray, Ethiopia, 2015. BMC Res Notes. 2018 May 24;11(1):339. doi: 10.1186/s13104-018-3432-4. PMID 29793551
- [Background] Khilnani P, Sarma D, Singh R, Uttam R, Rajdev S, Makkar A, Kaur J. Demographic profile and outcome analysis of a tertiary level pediatric intensive care unit. Indian J Pediatr. 2004 Jul;71(7):587-91. doi: 10.1007/BF02724117. PMID 15280607